CLINICAL TRIAL: NCT02140697
Title: Efficacy and Safety of Hippophae Rhamnoides L. Leaf Extract on Body Fat
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SS-BF-HLE
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hippophae rhamnoides L. Leaf Extract (Experimental): Hippophae rhamnoides L. Leaf Extract 3g/day
  Interventions: Dietary Supplement: Hippophae rhamnoides L. Leaf Extract (3g/day)
- Placebo (Placebo Comparator): Placebo 3g/day
  Interventions: Dietary Supplement: Placebo (3g/day)

INTERVENTIONS:
Dietary Supplement: Hippophae rhamnoides L. Leaf Extract (3g/day) — Hippophae rhamnoides L. Leaf extract (3g/day), parallel design
  Arms: Hippophae rhamnoides L. Leaf Extract
Dietary Supplement: Placebo (3g/day) — Placebo (3g/day), parallel design
  Arms: Placebo

SUMMARY:
Obesity is a major health issue worldwide; there is a constant raise in obesity related death each year. In vitro and animal studies elucidated Hippophae rhamnoides L. Leaf Extract as a novel anti-obesity agent. However, the efficacy and safety of Hippophae rhamnoides L. Leaf Extract supplementation on body weight regulation in humans are lacking.

DETAILED DESCRIPTION:
The investigators performed a 12-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Hippophae rhamnoides L. Leaf Extract on body fat. The investigators measured Body Fat Mass, Percent Body Fat, Fat Free Mass, weight, and body mass index.

ELIGIBILITY:
Inclusion Criteria:

* age between 19 and 65 years,
* BMI 25~29.9 kg/m2 or Waist circumference ≥ 90(men), ≥ 85(women),
* subjects giving written informed consent

Exclusion Criteria:

* BMI ≥ 30 kg/m2
* Significant variation in weight(more 10%) in the past 3 months
* Cardiovascular disease, e.g. arrhythmia, heart failure, myocardial infarction, and patient with pacemaker
* History of disease that could interfere with the test products or impede their absorption, such as gastrointestinal disease or gastrointestinal surgery
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnancy or breast feeding etc,.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in body fat mass | Baseline and 12 week
  Body fat mass was measured in study baseline and visit 3(12 week).

SECONDARY OUTCOMES:
Change in percent body fat | Baseline and 12 week
  Percent body fat was measured in study baseline and visit 3(12 week).
Change in fat free mass | Baseline and 12 week
  Fat Free Mass was measured in study baseline and visit 3(12 week).
Change in weight | Baseline and 12 week
  Weight was measured in study baseline and visit 3(12 week).
Change in body mass index | Baseline and 12 week
  Body mass index was measured in study baseline and visit 3(12 week).

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea